CLINICAL TRIAL: NCT05911906
Title: An Open-label, Clinical Feasibility Study of the Efficacy of Remdesivir for Long-COVID.
Acronym: ERASE-LC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Derby (Other)
Collaborators: University of Exeter (Other); University of Plymouth (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other); Aston University (Other); Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark Faghy, Professor in Clinical Exercise Science, University of Derby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UoD/ERASE-LC/23
Record Dates: First submitted 2023-06-20; First posted 2023-06-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Long COVID; Anti-virals; Remdesivir; Long COVID Symptoms
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: One study group will receive Remdesivir.
Masking Description: Open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Five days of Remdesivir infusion delivered by IV.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — Remdesivir is a prodrug that is intended to allow intracellular delivery of GS-441524 monophosphate and subsequent biotransformation into GS-441524 triphosphate, a ribonucleotide analogue inhibitor of viral RNA polymerase.
  Participants will receive a single loading dose of 200 milligrams of Remdesivir in 250ml sodium chloride 0.9% bag via IV over 60 minutes on day 1, followed by, on days 2 - 5, a dose of 100 milligrams of Remdesivir in 250ml sodium chloride 0.9% bag via IV once daily over 30 minutes.
  Other Names: Veklury; PRD8099279

SUMMARY:
Following an infection with Severe Acute Respiratory Syndrome coronavirus 2 (SARS-CoV2), one in ten people will experience persisting symptoms, or develop symptoms which can last for months and even years. These symptoms affect people in different ways and have been demonstrated to broadly impact physical, mental, and cognitive health. This is called Long COVID. Currently, there are no treatments available to address the issues that patients experience but anti-viral medications have been suggested as being potentially effective. This study will recruit patients that have confirmed long COVID and participants will undertake a series of tests to determine their symptoms and the impact that their condition has had on their bodily systems. The total duration of each participant's involvement is approximately 8 weeks, and this will involve 13 visits (15 visits if taking part in Exeter) at the closest study location (Derby or Exeter). Initial assessments are conducted over three separate visits and then all participants will be scheduled to receive five consecutive days of a medication that has been identified as having the potential to reduce the impact of Long COVID. Following a period of 28 days, participants will be invited to repeat the same tests that were conducted before receiving the medication so that it can be determined how well the drug has worked. In this study we are specifically collecting information to understand how feasible this medication could be to help patients improve their condition and this will help us to determine how likely this drug is able to be used within the wider Long COVID community.

The medication that will be used within this study is an existing anti-viral medication (Remdesivir). If we find patients are able to tolerate the treatment and the research tasks we will use this information to conduct a larger trial to determine how well this drug can be used to reduce the impact of Long COVID in a greater number of patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of enrolment
* Previously confirmed or suspected SARS-CoV-2 infection
* Confirmed diagnosis of Long COVID by a Health Care Practitioner according to the *definition provided by the World Health Organisation for persistent symptoms following a confirmed SARS-CoV-2 infection.
* Willing and able to provide informed consent, complete the surveys, and complete all planned clinical assessments, and return for scheduled study visits.
* Evidence of persistent symptom profile relative to pre-COVID-19 status as derived from patient reported outcome measures.
* Lives within commutable distance of the relevant centre, at discretion of local Principal Investigator.

  * WHO define Long COVID as the continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation.

Exclusion Criteria:

* Treatment history of Remdesivir, molnupiravir, paxlovid and/or any other COVID-19 anti-viral medication (<6 months).
* A diagnosis of a compromised immune system or function from a Healthcare Professional.
* Currently engaged in a physical rehabilitation programme or intervention aimed to improve Long COVID symptom profile and/or functional status.
* Recognised as a 'severe risk' of experiencing post-exertional malaise following engagement in physical tasks. Determined using the Modified De Paul Symptom Questionnaire.
* Lack of mental capacity to provide informed consent.
* Unable to understand verbal English/have a hearing impairment that prevents adequate communication.*
* Participation in another clinical drugs trial within the last 6 months
* Currently pregnant, breastfeeding or attempting to get pregnant (i.e., not using effective methods of contraception).
* Currently taking medications known to have an interaction with Remdesivir (e.g., chloroquine phosphate or hydroxychloroquine) as defined by British National Formulary (BNF) information on the selection, prescribing, dispensing and administration of medicines: https://bnf.nice.org.uk/interactions/Remdesivir/
* History of serious adverse reactions to anti-viral medication and intravenous infusions
* History of Hepatic or Renal Impairment (eGFR (<30ml/min) and LFTs ALT>x5 ULN).
* Exeter participants only: No recent/long standing history of CT (within 3 months)/ ongoing radiotherapy treatment. Risks of accumulative burden to be discussed as part of study involvement but it is at the discretion of participants.

  *Note:
* English Comprehension: Potential participants who are unable to understand verbal English will not be eligible for this study. This is due to the necessity of telephone contact which is a key aspect of this study and the unavailability of validated questionnaires in languages other than English.
* Hearing Impairment: Unfortunately, if the participant has a hearing impairment that prevents adequate communication on the telephone, they will not be able to take part in the study. This will be clearly stated in the participant information sheet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  To ascertain screening and recruitment rates (overall and by different recruitment pathways).
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  Retention and dropout rate (due to the treatment and/or trial demands, overall and by centre):
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 22 days
  Adherence to treatment regimen (attendance to 5 days of IMP).
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  Completeness of study assessments (CPET, Bloods and PET/CT if in Exeter).
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  Completeness of all data collection activities including baseline and +28 days after treatment.
To assess the feasibility of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  Acceptability of outcome measurements (measured by completion rates).

SECONDARY OUTCOMES:
To identify the most clinically relevant primary outcome for the definitive study | 52 days
  Quality of life, functional status and symptom burden (Pre and Post Intervention Patient Reported Outcome Measures)
To identify the most clinically relevant primary outcome for the definitive study | 52 days
  Tolerance to physical stimulus: exercise tolerance and reduced post exertional symptom exacerbation following incremental exercise.
To identify the most clinically relevant primary outcome for the definitive study | 52 days
  Physiological function, physical function, cognitive function, and emotional status and/or capacity.
To identify the most clinically relevant primary outcome for the definitive study | 52 days
  Biomarker and inflammatory profiles
To identify the most clinically relevant primary outcome for the definitive study | 55 days
  Exeter patients only - Microvascular function: whole body FDG uptake using PET/CT methods.
To determine the clinical safety and tolerance parameters of the use of Remdesivir in the treatment of patients with Long COVID. | 55 days
  AE/SAE/AR/SAR/SUSAR

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Allgar, PhD, Study Chair — Pen CTU
Locations (4):
- United Kingdom (4):
  - University of Derby, Derby, Derby
  - Derbyshire Community Health Services NHS Foundation Trust, Chesterfield
  - Royal Derby Hospital (UHDB), Derby
  - University of Exeter / Royal Devon University Healthcare NHS FT, Exeter

IPD SHARING:
Plan to Share IPD: Yes
The PenCTU data team will have access to the trial dataset, including identifiable participant data. Other members of the CTU and the wider study team will have restricted access to pseudo-anonymised study data. Access to the dataset will be granted to the Sponsor and host institution on request, to permit study-related monitoring, audits and inspections. Access will be overseen by the CTU data manager and trial manager. Access to the final dataset will be provided to the trial statisticians for analysis. After the trial has been reported, the anonymised individual participant data that underlie the results will be available on request from the CI and Sponsor, along with supplementary files as required (e.g., data dictionaries, blank data collection forms, analysis code, etc). Data will be shared with (or access to the data will be provided to) requestors whose proposed use of the data has been approved by the CI and Sponsor, under an appropriate data-sharing agreement.

REFERENCES:
- See also: Study website — https://www.plymouth.ac.uk/research/penctu/erase-long-covid